CLINICAL TRIAL: NCT05063617
Title: Assessing the Acceptability and Feasibility of an mHealth App to Increase the Quantity and Quality of Physical Activity Experiences Among Individuals With Spinal Cord Injury Who Ambulate
Brief Title: SCI Step Together: Improving Physical Activity Participation Among Individuals With SCI Who Ambulate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Curatio Networks Inc. (Unknown)
Responsible Party: Principal Investigator, Kathleen Martin Ginis, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCIStepTogether; H21-01279 (Other: UBC)
Record Dates: First submitted 2021-08-10; First posted 2021-10-01 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Spinal Cord Injuries
Keywords: exercise; health promotion; smartphone; telemedicine; recreation
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either a wait-list control or intervention group. The wait-list control group will be instructed to maintain their current health habits and not to engage in any new physical activity or health programs for the next 8-weeks. The wait-list control group will be invited to access the intervention after 8-weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-List Control (No Intervention): The wait-list control group will be instructed to maintain their current health habits and not to engage in any new physical activity or health programs for the next 8-weeks. The wait-list control group will be invited to access the intervention after 8-weeks.
- mHealth Intervention (Experimental): Intervention participants will be directed to the App store to download the Stronger Together app to proceed with app registration. Participants will then be connected with the community coach who is a 'real live person' who monitors in-app activity (this will be the program lead, SL). Other in-app features include peer discussion groups, behavioural support, and educational modules to support strategies to increase the quantity and quality of physical activity.
  Interventions: Device: SCI Step Together

INTERVENTIONS:
Device: SCI Step Together — The 8-week program features weekly blocks of content. Each week builds from the previous week and targets specific components related to the three basic psychological needs (autonomy, relatedness, competence). The overall cadence of each weekly block is maintained throughout. For example, each week contains: 1) education modules 2) a worksheet or guided practice to apply the strategies in their own goals for that week along with embedded questions to discuss with their community coach 3) behavioural support from the community coach and 4) peer support from the discussion group.
  Arms: mHealth Intervention

SUMMARY:
The project aims to test the feasibility of a new digital (mHealth) physical activity support program, delivered through an innovative mHealth platform (Curatio) for individuals living with spinal cord injury (SCI) who walk. The rationale for this project is to understand whether a mHealth intervention for increasing the amount and quality of physical activity is feasible for individuals with SCI who walk. The plan is to assess engagement, acceptability and feasibility in addition to primary outcomes related to physical activity behaviour. The investigators hypothesize that the intervention will be feasible and acceptable to deliver to individuals with SCI who walk. The investigators also hypothesize that the intervention will be engaging but recommendations will be made by participants following the study. Finally, it is hypothesized that compared with individuals in the wait-list control group, individuals in the intervention group will experience the following improvements related to exercise after 8-weeks: fulfillment of basic psychological needs, greater autonomous motivation, have enhanced social support, better action control, improved facilitators for behaviour change, more leisure-time physical activity, better quality participation, and enhanced employment.

DETAILED DESCRIPTION:
This randomized controlled trial will examine the feasibility and acceptability of a mobile health (mHealth) application called Stronger Together. Stronger Together is an app that hosts programs for individuals with chronic illnesses and disabilities. In this study, the investigators are developing and testing the Stronger Together program that aims to improve the quantity and quality of physical activity among ambulators with SCI. Furthermore, the study will also collect pilot data on the magnitude of the effects on physical activity participation (quality and quantity) and psychosocial influences on physical activity. Individuals living with SCI who walk and live in Canada or the United States will be recruited for this study and will be assigned to either a wait-list control or intervention group. The wait-list control group will be instructed to maintain current health habits and not to engage in any new physical activity or health programs for the next 8-weeks. The wait-list control group will be invited to access the intervention after 8-weeks.

Potential participants will be immediately directed to complete the consent forms/baseline measures in Qualtrics. Once consent and baseline measures are completed, participants will be randomized into either the wait-list control or intervention condition. The investigators will aim to recruit at least 8-10 participants with consent and baseline measures completed before randomization into conditions in order for there to be enough participants in the program at the same time for peer support. After the first 8-10 participants, individuals will be randomized immediately after baseline testing so that participants randomized to the intervention group can join others in the app right away. Randomization will be done by the investigators using a random numbers generator in blocks of 2 and 4 with even groups in each condition (i.e., n=10 per condition). Waitlist-control participants will be directed to continue normal daily activity. Intervention participants will be directed to the App store to download the Stronger Together app to proceed with app registration. Participants will then be connected with the community coach who is a 'real live person' who monitors in-app activity. Other in-app features include peer discussion groups, behavioural support, and educational modules to support strategies to increase the quantity and quality of physical activity.

The 8-week program features weekly blocks of content. Each week builds from the previous week and targets specific components related to the three basic psychological needs (autonomy, relatedness, competence). The overall cadence of each weekly block is maintained throughout. For example, each week contains: 1) education modules 2) a worksheet or guided practice 3) behavioural support from the community coach and 4) peer support from the discussion group. Participants in the intervention group will be encouraged to use the app as often as needed (but at least once per week) and actively participate in the programming. The community coach (SL) will prompt participants who have not engaged in the app in a week to remind participants to complete weekly modules. In-app data, including user metrics will be collected and analyzed for descriptive patterns and assess correlations with the outcome measures (e.g., is the amount of time spent in-app correlated with changes in behaviour).

Participants in both the intervention and control groups will be asked to participate in eight online questionnaires provided through the survey platform Qualtrics at three different time points (baseline/onboarding, 4- and 8-weeks of using the Stronger Together program). A link to these questionnaires which will be hosted on Qualtrics will be emailed to all participants.

After completing the final online survey (at 8-weeks), participants in the intervention group will be invited to participate in an interview to further explore their experiences and to increase understanding of factors that influence acceptability and satisfaction of the Stronger Together program. The interview will be structured whereby the participant will go through the application with the interviewer to discuss preferred components. This will provide a greater understanding of user engagement.

Additionally, feasibility metrics will be kept and recorded throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Can read and write in English
* Own a smartphone or tablet
* Are 19 years of age or older
* Are a Canadian or United States resident
* Have sustained a spinal cord injury
* Walk for their daily mode of mobility

Exclusion Criteria:

* Have a spinal cord injury but use a wheelchair as primary mode of mobility

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 8 weeks
  Divide the total number of participants enrolled by the number of participants contacted
Eligibility rate | 8 weeks
  Number of potential participants excluded from the total number of interested participants
Retention rate | 8 weeks
  Number of participants who completed at least some part of the intervention from those who were randomized
Adherence rate | 8 weeks
  Number of participants who completed testing and follow-up measures
Costs | 8 weeks
  Cost of producing software and app, participant remuneration, and cost of health behaviour coach
Staff preparation time | Feasibility metrics will be recorded throughout the study. Feasibility will be assessed at the end of the 8-weeks.
  The number of hours it requires staff to recruit partners and participants, liaise participants, and enter participant data
Number of adverse events | 8 weeks
  Number of health problems reported over the course of the intervention
Compliance | 8 weeks
  The number of modules completed by each intervention participant in the app
Number of log ins | 8 weeks
  The number of times each intervention group participant logs into the app on a weekly basis
Duration of log ins | 8 weeks
  The duration of each log in for each intervention group participant on a weekly basis
Qualitative interview | 8 weeks
  A semi-structured interview with intervention group participants to explore the experiences with the app
Basic Psychological Needs - The Psychological Need Satisfaction in Exercise Scale. | Change in Basic Psychological Needs will be assessed at three time points: Baseline, Week 4, and Week 8
  Basic Psychological Needs will be assessed using the The Psychological Need Satisfaction in Exercise Scale (Wilson et al., 2006). This 18-item scale assesses the satisfaction of the psychological needs for exercise using a 6-point Likert scale ranging from 1 (false) to 6 (true) (Wilson et al., 2006). A mean can be calculated for each psychological need (6-items each for autonomy, competence, and relatedness) with a higher score representing greater satisfaction of that need.
Social Support - Sallis' social support questionnaire | Change in Social Support will be assessed at three time points: Baseline, Week 4, and Week 8
  Social support will be measured using a modified version of Sallis' social support questionnaire (Sallis et al., 1987). The 7-item survey uses a 6-point Likert-type scale and assesses emotional support (3 items) and practical support (4 items). A higher score means individuals feel a greater sense of social support.
Autonomous and Controlled Motivation - The Treatment Self-Regulation for Exercise Scale | Change in Motivation will be assessed at three time points: Baseline, Week 4, and Week 8
  Motivation will be assessed by the The Treatment Self-Regulation for Exercise Scale. The 15-item scale uses a 7-point Likert scale ranging from 1 (not at all true) to 7 (very true) to assess why one would engage in exercise activities (Levesque et al., 2007). A higher score is more autonomous motivation.
Behaviour Change Factors - The Determinants of Physical Activity Questionnaire | Change in Behaviour Change Factors will be assessed at three time points: Baseline, Week 4, and Week 8
  Behaviour change factors will be assessed using the The Determinants of Physical Activity Questionnaire. A modified version will be used to assess the following domains targeted in the intervention: Knowledge, Beliefs about Capabilities, Skills, Social Influences, Beliefs about Consequences, Action Planning, Coping Planning, and Goal Conflict (24-items). The questionnaire uses a scale from 1 to 7 with 1 being strongly disagree, and 7 being strongly agree.
Action Control - The Action Control Scale (Sniehotta et al., 2005). | Change in Action Control will be assessed at three time points: Baseline, Week 4, and Week 8
  Action control will be assessed with 6 items that ask participants to indicate the extent to which they self-monitor their physical activity (1 = definitely false; 7 = definitely true). (Sniehotta et al., 2005).

SECONDARY OUTCOMES:
Leisure-Time Physical Activity - The Leisure-Time Physical Activity Questionnaire | Change in Leisure-Time Physical Activity will be assessed at three time points: Baseline, Week 4, and Week 8
  Physical activity will be measured using the The Leisure-Time Physical Activity Questionnaire-SCI (LTPAQ-SCI).
Quality of Physical Activity Participation - Measure of Experiential Aspects of Participation | Change in Quality of Physical Activity Participation will be assessed at three time points: Baseline, Week 4, and Week 8
  Quality of physical activity participation will be assessed using The Measure of Experiential Aspects of Participation (MeEAP).The scale is a questionnaire to assess the six experiential aspects of participation (i.e., belongingness, meaning, mastery, engagement, challenge, and autonomy) across life domains (Caron et al., 2019). The scale is completed separately for each life domain with 12-items. Participants will be asked to complete the scale for the exercise and sport domains only, for a total 24 items. Participants respond using a 7-point Likert type scale ranging from 1 (strongly disagree) and 7 (strongly agree).
Employment - The Short Form Craig Handicap Assessment and Reporting | Change in Employment will be assessed at three time points: Baseline, Week 4, and Week 8
  Employment will be assessed using the Craig Handicap Assessment and Reporting Technique - Short Form (CHART-SF).The CHART-SF will be modified to 2-items for the current study to only assess employment hours and financial earnings.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Martin Ginis, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Sharing individual participant data is not part of our ethical approval.

REFERENCES:
- [Derived] Lawrason SVC, Brown-Ganzert L, Campeau L, MacInnes M, Wilkins CJ, Martin Ginis KA. mHealth Physical Activity Intervention for Individuals With Spinal Cord Injury: Planning and Development Processes. JMIR Form Res. 2022 Aug 19;6(8):e34303. doi: 10.2196/34303. PMID 35984695

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT05063617/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT05063617/ICF_001.pdf